CLINICAL TRIAL: NCT00003475
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients With Primary Malignant Brain Tumors
Brief Title: Antineoplaston Therapy in Treating Patients With Primary Malignant Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066512; BC-BT-21 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Malignant Brain Tumors
Keywords: adult glioblastoma multiforme; adult anaplastic astrocytoma; adult anaplastic astrocytoma/Mixed
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a primary malignant brain tumor that has not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adults with primary malignant brain tumors that have not responded to standard therapy provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adults with primary malignant brain tumors that have not responded to standard therapy.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with primary malignant brain tumors that have not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with primary malignant brain tumors that have not responded to standard therapy, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with a primary malignant brain tumor.

OVERVIEW: This is a single arm, open-label study in which adults with malignant brain tumors that have not responded to standard therapy receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed incurable adult primary malignant brain tumor
* Evidence of progressive or recurrent tumor by MRI scan performed within 2 weeks prior to study entry
* Must have received and failed standard therapy
* Tumor must be at least 5 mm
* No brain stem tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* Hematological function normal
* WBC at least 2000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* No liver failure
* No evidence of hepatic insufficiency
* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal

Renal:

* No evidence of renal insufficiency
* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No chronic heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease, such as severe chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No medical or psychiatric illness that would preclude study treatment
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy, except in patients with disease progression during initial therapy
* At least 6 weeks since prior nitrosoureas, except in patients with disease progression during initial therapy
* No concurrent antineoplastic agents

Endocrine therapy:

* Corticosteroids allowed

Radiotherapy:

* See Disease Characteristics
* At least 8 weeks since prior radiotherapy, except in patients with disease progression during initial therapy

Surgery:

* At least 4 weeks since prior surgery, except in patients with disease progression during initial therapy

Other:

* Recovered from prior therapy
* Cytodifferentiating agents allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski SR, Janicki TJ, Burzynski GS. A phase II study of antineoplastons A10 and AS2-1 in adult patients with recurrent glioblastoma multiforme: Final report (protocol BT-21). Journal of Cancer Therapy 5:946-956, 2014. DOI: http://dx.doi.org/10.4236/jct.2014.510100
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourty patients were recruited between February 1996 and February 2011. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therpay: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a primary malignant brain tumor that has not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
Period: Overall Study
Arm/Group | Antineoplaston Therpay
Started | 40
Completed | 27
Not Completed | 13
Not completed — Not evaluable | 13

BASELINE CHARACTERISTICS:
Groups:
- Antineoplaston Therpay: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Adults with a primary malignant brain tumor that has not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
Arm/Group | Antineoplaston Therpay
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 48.2 [19.7 to 68.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Groups:
- Antineoplaston Therpay: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a primary malignant brain tumor that has not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Arm/Group | Antineoplaston Therpay
Number analyzed (Participants) | 27
Participants
  Complete Response | 2
  Partial Response | 2
  Stable Disease | 4
  Progressive Disease | 19

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therpay
Number analyzed (Participants) | 40
Percentage of participants
  6 months overall survival | 47.5
  12 months overall survival | 27.5
  24 months overall survival | 2.5
  36 months overall survival | 2.5
  48 months overall survival | 2.5
  60 months overall survival | 2.5

ADVERSE EVENTS:
Time Frame: 15 years, 2 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a primary malignant brain tumor that has not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 21/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 1 — The Hemoglobin was not related to Antineoplaston therapy.
Central venous catheter infection (Infections and infestations) | 2 — The Central venous catheter infections were not related to Antineoplaston therapy.
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1 — The Pancreatic endocrine: glucose intolerance was not related to Antineoplaston therapy.
Perforation, GI: Colon (Gastrointestinal disorders) | 1 — The Perforation, GI: Colon was not related to Antineoplaston therapy.
Infection - Other (Infections and infestations) | 1 — The Infection - Other was not related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 4 — The Infections (documented clinically): Lung (pneumonias) were not related to Antineoplaston therapy.
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 1 — The Infection (documented clinically): Skin (cellulitis) was not related to Antineoplaston therapy.
Mood alteration: Agitation (Nervous system disorders) | 1 — The Mood alteration: Agitation was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 5 — The Seizures were not related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 5 — The Somnolences/depressed levels of consciousness were not related to Antineoplaston therapy.
Pain: Back (Musculoskeletal and connective tissue disorders) | 1 — The Pain: Back was not related to Antineoplaston therapy.
Pain: Head/headache (Nervous system disorders) | 2 — The Pain: Head/headaches were not related to Antineoplaston therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 — The Dyspnea (shortness of breath) was not related to Antineoplaston therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 3 — The Thromboses/thrombi/embolisms were not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 8
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 10
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 7
Hypertension (Cardiac disorders) | 3
Central venous catheter infection (Infections and infestations) | 5
Non-functional central venous catheter (General disorders) | 7
Central venous catheter - Other (General disorders) | 5
PT (Blood and lymphatic system disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 20
Fever (General disorders) | 6
Rigors/chills (General disorders) | 3
Edema/Fluid retention (General disorders) | 15
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 5
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 11
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 12
Hemorrhage, GU (Renal and urinary disorders) | 3
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 3
Infection - Other (Infections and infestations) | 4
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 6
Infection (documented clinically): Mucosa (Infections and infestations) | 5
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 4
Opportunistic infection (Infections and infestations) | 3
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3
Hypercholesteremia (Investigations) | 4
Hyperglycemia (Investigations) | 17
Hypernatremia (Investigations) | 24
Hypocalcemia (Investigations) | 12
Hypoglycemia (Investigations) | 7
Hypokalemia (Investigations) | 30
Hypophosphatemia (Investigations) | 6
Metabolic/Laboratory - Other (Investigations) | 3
Proteinuria (Investigations) | 4
SGOT (Investigations) | 6
SGPT (Investigations) | 8
Uric acid, serum-high (hyperuricemia) (Investigations) | 3
Ataxia (incoordination) (Nervous system disorders) | 6
Confusion (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 10
Memory impairment (Nervous system disorders) | 4
Mood alteration: Depression (Nervous system disorders) | 3
Neuropathy: motor (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 11
Somnolence/depressed level of consciousness (Nervous system disorders) | 20
Speech impairment (Nervous system disorders) | 5
Vision-blurred vision (Eye disorders) | 3
Pain: Back (Musculoskeletal and connective tissue disorders) | 3
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 4
Pain: Head/headache (Nervous system disorders) | 15
Pain: Joint (Musculoskeletal and connective tissue disorders) | 4
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Urinary frequency/urgency (Renal and urinary disorders) | 5
Thrombosis/thrombus/embolism (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No